CLINICAL TRIAL: NCT04554992
Title: Convalescent Plasma for the Treatment of Coronavirus Disease 2019
Brief Title: Convalescent Plasma for the Treatment of COVID-19 (Coronavirus Disease 2019)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Eric Salazar, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00025121
Record Dates: First submitted 2020-08-26; First posted 2020-09-18 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Given that this is a pilot study to evaluate the safety of treatment with convalescent COVID-19 plasma versus standard care in subjects with severe and/or critical COVID-19 between the cases and historical controls without predetermined data, a convenient sample size of 700 patients (350 per group) has been proposed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All subjects recruited will be transfused with COVID 19 convalescent plasma. A prospective comparison with matched historical controls receiving standard care will be employed.
  Interventions: Biological: COVID 19 Convalescent Plasma

INTERVENTIONS:
Biological: COVID 19 Convalescent Plasma — COVID 19 convalescent plasma is a blood product collected from donors who have recovered from a previous COVID 19 infection

SUMMARY:
This pilot, prospective study will assess the safety and efficacy of COVID-19 convalescent plasma versus standard care as treatment for severe and/or critical COVID-19 (as defined in the inclusion criteria) in adults 18 years of age and older. A total of 350 eligible subjects will receive a transfusion of anti-SARS-CoV2 ( severe acute respiratory syndrome) convalescent plasma.

DETAILED DESCRIPTION:
Patients meeting inclusion/exclusion criteria will be approached for study consent based on the time of hospital admission and the availability of an blood type compatible product. 300mL plasma units of COVID-19 convalescent patients will be utilized for transfusion. During a period of 14 days, the patient will be eligible to receive up to 10 units of plasma, to be completed with 4 hours as per institutional transfusion standard operating procedures. Transfusion by apheresis (plasma exchange) may be employed to reduce the risk of volume overload. The number of units to be used will be determined by the study team based on protocol inclusion and exclusion criteria, and clinical evaluation of the patient's severity and response.

Subjects will be followed for at least 60 days or up to 3 months following initial transfusion for adverse event monitoring and data collection.

ELIGIBILITY:
Inclusion Criteria:

Recipient must meet criteria outlined in the recent Investigational COVID-19 Convalescent Plasma - Emergency INDs (investigational new drug) guidance (https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds)

Exclusion Criteria:

1. History of prior severe reactions to transfusion of blood products with imputability of probable or definite as defined by Center of Disease Control National Healthcare Safety Network Hemovigilance Module [see https://www.cdc.gov/nhsn/PDFs/Biovigilance/BV-HV-protocol-current.pdf].
2. Has underlying uncompensated and untreatable end stage disease.
3. Fluid overload or other condition that would contraindicate administration of plasma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of serious adverse events related to the treatment intervention. | up to 60 days post-transfusion
  Total number of grade 3 and above throughout study period
Mortality at Day 28 post-hospital admission. | up to 28 days post-transfusion
  All cause mortality at day 28

SECONDARY OUTCOMES:
Length of hospital stay | up to 60 days post-transfusion
  Total number of days subjects are hospitalized during study period
Length of supplemental oxygen requirement. | up to 60 days post-transfusion
  Total number of days subjects requires supplemental oxygen during study period
Length of mechanical ventilation requirement. | up to 60 days post-transfusion
  Total number of days subjects require mechanical ventilation during study period
Length of ICU stay | up to 60 days post-transfusion
  Total number of days subject is subject stays in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Eric Salazar, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hopsital, Houston, Texas, United States